CLINICAL TRIAL: NCT00159354
Title: Evaluation of Smoking-Induced Neutrophil Activation as a Potential Biomarker of Response to Therapeutic Interventions in COPD: Proof of Concept Study
Brief Title: Measurement of Smoking-Induced Neutrophil Activation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDG-PETsmoking
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: COPD
Keywords: FDG-PET; pulmonary inflammation,; smoking,; COPD; steroid intervention
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Pneumonia; Smoking

INTERVENTIONS:
Drug: predisolone

SUMMARY:
Neutrophil involvement in the development of COPD by smokers is well recognised. However not all smokers develop overt lung disease. We have previously shown that uptake of FDG is related to neutrophil activity and can be measured by PET and that uptake is greater in COPD patients than normal subjects. We have also shown that FDG-PET shows inflammatory changes in asymptomatic smokers after cigarette smoking. We plan to investigate the attenuation of this inflammation by steroid tablets and whether FDG PET can demonstrate this. We also wish to establish if similar changes are demonstrated after smoking by COPD patients.

DETAILED DESCRIPTION:
Asymptomatic smokers will be recruited by advertisement in newspapers and from posters displayed in the local community.Patients will be recruited from Hammersmith Hospital NHS Trust and local GP surgeries, where we shall display posters. We shall also directly ask patients whom we think may be suitable. This could be at a respiratory clinic, after they attend the lung function department for routine tests, and at GP and practice nurse appointments. After discussing the research outline with the subjects, either in person or by phone, we shall give them the information sheet and ask them to attend for a screening visit. This will be a chance for them to ask more questions, and for us to obtain informed consent. We will then carry out a brief medical examination and routine lung function tests. Providing they fulfil the inclusion criteria we shall then organise the subsequent visits, for 2 scans if they are patients with COPD or 3 if they are asymptomatic smokers. All participants will undergo chest X-ray to exclude other lung disease, unless they have had one in the past year. They must abstain for smoking for at least 12 hours prior to visit, and fast for 4 hours prior to scan. On the first day of attendance they will have a brief medical to assess whether they are clinically stable, and have spirometry and CO monitored, to confirm abstinence. For the scan visits the asymptomatic smokers will take the placebo or prednisolone the previous evening at 10pm and again the next morning with a light breakfast by 7:30am. On 2 scan days they will smoke 2 cigarettes 4h later, 60 minutes prior to scan. The PET scan takes about 90 minutes, and includes blood sampling throughout. They must be able to lie still in the scanner. We will aim to complete the scans at 1-2 week intervals, whilst clinically stable.

The COPD patients will not take prednisolone/placebo, but will either smoke 2 real or dummy cigarettes prior to scan. This protocol is similar to others used previously, which have proved acceptable to COPD patients and healthy smokers.

ELIGIBILITY:
Inclusion Criteria:

* Male smokers >10 pack.year history,
* FEV1>80% predicted,
* no relevant medical or mental disorder, able to give informed consent and
* Patients with COPD,
* >20 pack.year history,
* no other active lung disease,
* FEV1<70%
* FEV1/VC<70%,
* no other relevant medical or mental disorder, able to give informed consent

Exclusion Criteria:

* Female asymptomatic smokers
* ex-smokers
* other lung disorder
* relevant medical or mental illness
* recent (within 1 month) chest infection
* diabetes

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2005-06; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Modification of neutrophil activation

CONTACTS AND LOCATIONS:
Overall Officials: Hazel A Jones, PhD, Principal Investigator — Imperial College London
Locations (1):
- Hammersmith Campus, London, United Kingdom